CLINICAL TRIAL: NCT02939521
Title: Reconstructive Surgical Approach for Pincer Nail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica María del Mar Ruiz (Other)
Responsible Party: Principal Investigator, MARIA DEL MAR RUIZ HERRERA, Director, Clínica María del Mar Ruiz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Maria del Mar Ruiz-Herrera
Record Dates: First submitted 2016-10-12; First posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Pincer Nail
Keywords: Pincer Nail; Surgery
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental): Consists of a dorsal flattening of of the bone at the distal phalanx, with a frontal lifting of the distal skin of the toe
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery

SUMMARY:
A prospective design that studies the effects of a new technique for the treatment of pincer nails. The technique consists of a flattening of the bone of the distal phalanx with a frontal skin lifting that is performed in patients with a pincer nail deformity. Visual Analog Scale (VAS) will be measure before surgery, one month and one year after surgery.

ELIGIBILITY:
Eligibility Criteria:

* Pincer nail deformity
* At least 5 years of pain in the nail
* Prior unsuccessful conservative treatments

Exclusion Criteria:

* Medical or mental conditions that contraindicate surgical treatment of the condition.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Pain - 10 points Visual Analog Scale (VAS) | Change in Pain will be measured with a VAS: at baseline, after 1 month of treatment and after 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mª del Mar Ruíz-Herrera, DPM, Study Director — Mª del Mar Ruiz Clinic

IPD SHARING:
Plan to Share IPD: No